CLINICAL TRIAL: NCT02867384
Title: A Randomized Phase 2 Study of Obinutuzumab for Prevention of Chronic Graft-vs.-Host Disease After Allogeneic Peripheral Blood Stem Cell Transplantation
Brief Title: Obinutuzumab in cGVHD After Allogeneic Peripheral Blood Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Roche-Genentech (Industry)
Responsible Party: Principal Investigator, Corey S. Cutler, MD, MPH, MD, MPH, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-256
Record Dates: First submitted 2016-08-11; First posted 2016-08-15 (Estimated); Results first posted 2025-03-12 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Graft vs. Host Disease
Keywords: Graft vs. Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — obinutuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Obinutuzumab (Active Comparator): Obinutuzumab or will be administered at a pre- determine dose, intravenously, at 3, 6, 9 and 12 months from transplantation.
  * Premedication with histamine blockers and acetaminophen will be provided
  * All subjects will undergo allogeneic stem cell transplantation according to locally approved clinical trials
  Interventions: Drug: Obinutuzumab
- Placebo (Sham Comparator): Placebo will be administered at a pre- determine dose, intravenously, at 3, 6, 9 and 12 months from transplantation.
  * Premedication with histamine blockers and acetaminophen will be provided
  * All subjects will undergo allogeneic stem cell transplantation according to locally approved clinical trials
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Obinutuzumab — B cell depletion
  Other Names: Gazyva
  Arms: Obinutuzumab
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This research study is studying a drug called obinutuzumab as a means of preventing chronic Graft vs. Host Disease (cGVHD).

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease.

The FDA (the U.S. Food and Drug Administration) has not approved Obinutuzumab for prevention of chronic Graft-vs.-Host Disease (cGVHD), but it has been approved for other uses.

In this research study, the investigators are aiming to determine the effect of Obinutuzumab on the incidence of corticosteroid-requiring cGVHD after allogeneic Hematopoetic Cell Transplant (aHCT).

Chronic GVHD is a medical condition that can occur after bone marrow or stem cells are transplanted from one individual to another. After the transplant, the donor immune system may recognize the recipient body as foreign and may attempt to 'reject' the body. This process is referred to as Graft-vs. -Host Disease and may occur at any time, although generally not earlier than one hundred days after transplantation.

The immune system produces two types of lymphocytes (white blood cells), B cells and T cells. B cells are part of the 'memory' for the immune system, and they make antibodies (proteins) when bacteria, viruses or other potentially harmful materials enter the body. Obinutuzumab is an antibody, a molecule that targets certain cells by binding to specific parts of the target cell. In this case, Obinutuzumab will bind to a component of B cells called CD20, resulting in the B cell getting killed. It is thought that reducing the number of B cells will reduce the chances of developing cGVHD after transplant. Previous studies with another antibody targeting CD20 on B cells suggests that there may be a reduced chance of developing cGVHD and the need to prescribe Corticosteroids to treat cGVHD when B cells are killed.

This is a randomized, placebo controlled trial. This means that approximately half of the study participants will receive Obinutuzumab, and the other half will receive a placebo (saline solution). A computer will decide which participants will receive Obinutuzumab or placebo, and neither the participant or the study doctor will know which the participant has received until the study is completed. It is important to note that the current standard is to receive no therapy specifically to prevent cGVHD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects deemed potentially eligible by their treating physicians will be screened for enrollment after d+60 from transplantation
* Patients who have undergone either ablative or non-myeloablative allogeneic stem cell transplantation are eligible.
* Peripheral blood stem cells must have been used as the stem cell source.
* Patients must have received transplantation from donors (both related and unrelated) who are identical at 8 HLA loci (A, B, C and DR1), or mismatched at no more than 1 locus (7/8). Among related donors, HLA C typing is not required (6/6 HLA matches). Class I typing is to be performed by PCR-SSP techniques and CDC techniques. Class II typing is performed by PCR-RFLP +/- PCR-SSP techniques.
* No evidence of relapsed or residual malignancy within 30 days of trial entry. All patients must undergo appropriate staging for their malignancy (i.e. bone marrow aspiration for the Leukemias and PET-CT scanning for the lymphomas). Evidence of a persistent Cytogenetic abnormality will constitute evidence of residual or relapsed disease in the Leukemias, where present. Individuals with CLL are eligible if there is no more than 20% residual leukemia in the bone marrow at the time of study entry.
* Patients who have undergone a non-myeloablative stem cell transplant must have > 80% donor hematopoiesis within 30 days of study enrollment. Chimerism within 30 days of study entry must be greater than, equal to, or no more than 5% less than the chimerism measured at approximately day+30 (if performed).
* Age ≥ 18.0
* ECOG performance status ≤2 (Karnofsky ≥60%) (See Appendix A)
* Participants must have normal marrow function as defined by:

  * WBC ≥ 2,500/μL
  * Absolute Neutrophil Count ≥ 1,000/μL
  * Platelets ≥ 50,000/μL
* Ability to understand and the willingness to sign a written informed consent document.
* The effects of Obinutuzumab on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of Obinutuzumab administration.

Exclusion Criteria:

* Allogeneic stem cell transplantation using a single or multiple umbilical cord blood units or using bone marrow.
* Allogeneic stem cell transplantation using in vivo or ex vivo T cell depletion, either by cell manipulation or with T cell depleting antibodies (Any anti-thymocyte globulin preparation or alemtuzumab given within 30 days of transplantation)
* Participation in a clinical trial evaluating another preventative strategy for chronic GVHD, or ongoing participation in a clinical trial for therapy of acute GVHD. Prior completion of experimental therapy for acute GVHD is permissible if the experimental agent was used > 30 days prior to enrollment.
* Any evidence of ongoing gastrointestinal or hepatic acute GVHD, or evidence of greater than ongoing Stage I cutaneous acute GVHD. Ongoing, tapering therapy for resolved acute GVHD is permissible.
* Any evidence of prior active or resolved chronic GVHD.
* History of severe allergic reaction to Obinutuzumab
* No Donor Lymphocyte Infusion (DLI) prior to day 100, and no plans for a DLI in the upcoming 30 days.
* Evidence of any active uncontrolled infection (bacterial, viral or fungal) or evidence of natural exposure to Hepatitis B, Hepatitis C or HIV. Evidence of Hepatitis B exposure includes the presence of Hepatitis B surface antigenemia, a positive serological test for Hepatitis B core antibody or nucleic acid testing (NAT testing) that is positive for Hepatitis B. Vaccination to Hepatitis B is not an exclusion criteria.
* Pregnancy or lactation. Negative pregnancy test is required within the screening window
* Active use of any other investigational agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2024-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey Cutler, MD MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - Stanford University, Palo Alto, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Masonic Cancer Center, Minneapolis, Minnesota
  - Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 5 clinical sites in the U.S. from November 29, 2016 to January 30, 2023.
Groups:
- Obinutuzumab: Obinutuzumab will be administered at a pre- determine dose, intravenously, at 3, 6, 9 and 12 months from transplantation.
  * Premedication with histamine blockers and acetaminophen will be provided
  * All subjects will undergo allogeneic stem cell transplantation according to locally approved clinical trials
  Obinutuzumab: B cell depletion
- Placebo: Placebo will be administered at a pre- determine dose, intravenously, at 3, 6, 9 and 12 months from transplantation.
  * Premedication with histamine blockers and acetaminophen will be provided
  * All subjects will undergo allogeneic stem cell transplantation according to locally approved clinical trials
  Placebo: Placebo
- Never received treatment: Some patients never received any treatment and got randomized after enrollment.
Period: Overall Study
Arm/Group | Obinutuzumab | Placebo | Never received treatment
Started | 90 | 88 | 3
Randomized | 0 | 88 | 90
Completed | 39 | 30 | 0
Not Completed | 51 | 58 | 3
Not completed — GVHD requiring change in Treatment Medication | 14 | 30 | 0
Not completed — Progression/ Relapse | 15 | 19 | 0
Not completed — Adverse Event | 13 | 1 | 0
Not completed — Withdrawal by Subject | 6 | 5 | 0
Not completed — Physician Decision | 1 | 2 | 0
Not completed — Patient compliance | 1 | 0 | 0
Not completed — Intercurrent illness or uncontrolled infection | 1 | 1 | 0
Not completed — Never start treatment | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Obinutuzumab | Placebo | Never received treatment | Total
Number analyzed (Participants) | 90 | 88 | 3 | 181
Age, Continuous [Median (Full Range); unit: years] | 63 [21 to 79] | 63 [20 to 75] | 62 [39 to 63] | 63 [20 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 33 | 2 | 67
  Male | 58 | 55 | 1 | 114
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 76 | 79 | 2 | 157
  Black or African American | 3 | 2 | 0 | 5
  Asian | 0 | 2 | 0 | 2
  More Than One Race | 4 | 2 | 1 | 7
  Other | 7 | 3 | 0 | 10

OUTCOME MEASURES:

1. Primary Outcome: Rate Of Corticosteroid-Requiring cGVHD At One Year From HCT
Description: Percentage of participants who develop chronic Graft Versus Host Disease cGVHD requiring treatment with corticosteroids within the first year following Hematopoietic Cell Transplantation HCT.
Time Frame: 1 year
Population: The analysis only included patients who started treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Obinutuzumab: Obinutuzumab or will be administered at a pre- determine dose, intravenously, at 3, 6, 9 and 12 months from transplantation.
  * Premedication with histamine blockers and acetaminophen will be provided
  * All subjects will undergo allogeneic stem cell transplantation according to locally approved clinical trials
  Obinutuzumab: B cell depletion
Arm/Group | Obinutuzumab | Placebo
Number analyzed (Participants) | 90 | 88
percentage of participants | 13.3 [7.1 to 22.1] | 35.2 [25.3 to 46]
Statistical Analysis 1: Comparison: Obinutuzumab vs Placebo; Test type: Superiority; p = 0.0008, Fisher Exact

2. Secondary Outcome: Overall cGVHD Rate After HCT
Description: A secondary endpoint of this phase II trial is the overall rate cGVHD one and two years after HCT.
Time Frame: at 1 year and at 2 years
Reporting Status: Not Posted

3. Secondary Outcome: Immunosuppression-Free Survival (IFS) Rate
Description: IFS is defined as time from randomization to relapse, institution of systemic immune suppression, or death, whichever occurs first.
Time Frame: at 1 year and at 2 years
Reporting Status: Not Posted

4. Secondary Outcome: The Rate Of NIH Moderate-Severe cGVHD After HCT
Description: A secondary endpoint is the rate of NIH Moderate-Severe cGVHD one and two years after HCT.
Time Frame: at 1 year and at 2 years
Reporting Status: Not Posted

5. Secondary Outcome: Cumulative Incidence Of Non-Relapse Mortality And Relapse
Description: A secondary endpoint is the cumulative incidence of non-relapse mortality and relapse one and two years after HCT.
Time Frame: at 1 year and at 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were followed for 2 years. Deaths were monitored until 84.7 months.
Description: SAE is defined as an AE that results in: death or life-threatening illness; persistent or significant disability; a congenital anomaly/birth defect in an infant born to an Obinutuzumab-exposed mother or requires inpatient hospitalization or is considered a significant medical event by the investigator based on medical judgment. The analysis population is comprised of all randomized and treated patients. Only randomized and treated patients were monitored/assessed for AEs and All-Cause Mortality.
Arm/Group | Obinutuzumab | Placebo
All-Cause Mortality (participants affected / at risk) | 29/90 | 28/88
Serious Adverse Events (participants affected / at risk) | 28/90 | 12/88
Other Adverse Events (participants affected / at risk) | 87/90 | 81/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Obinutuzumab (N=90) | Placebo (N=88)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Heart failure (Cardiac disorders) | 1 | 0
Eye disorders - Other, specify (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 1
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0
Infusion related reaction (General disorders and administration site conditions) | 4 | 0
Lung infection (Infections and infestations) | 3 | 3
Sepsis (Infections and infestations) | 1 | 1
Upper respiratory infection (Infections and infestations) | 3 | 2
Infections and infestations - Other, specify (Infections and infestations) | 2 | 0
Neutrophil count decreased (Investigations) | 14 | 4
Platelet count decreased (Investigations) | 0 | 2
White blood cell decreased (Investigations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Visceral arterial ischemia (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Obinutuzumab (N=90) | Placebo (N=88)
Anemia (Blood and lymphatic system disorders) | 43 | 30
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 9 | 9
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 2
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 2 | 3
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 | 1
Hypoparathyroidism (Endocrine disorders) | 2 | 0
Hypothyroidism (Endocrine disorders) | 1 | 2
Blurred vision (Eye disorders) | 2 | 7
Cataract (Eye disorders) | 1 | 3
Dry eye (Eye disorders) | 16 | 34
Eye pain (Eye disorders) | 1 | 1
Flashing lights (Eye disorders) | 1 | 0
Floaters (Eye disorders) | 2 | 0
Papilledema (Eye disorders) | 0 | 2
Photophobia (Eye disorders) | 1 | 3
Scleral disorder (Eye disorders) | 0 | 2
Watering eyes (Eye disorders) | 1 | 0
Eye disorders - Other, specify (Eye disorders) | 3 | 5
Abdominal pain (Gastrointestinal disorders) | 6 | 8
Constipation (Gastrointestinal disorders) | 6 | 9
Diarrhea (Gastrointestinal disorders) | 24 | 16
Dry mouth (Gastrointestinal disorders) | 9 | 7
Dyspepsia (Gastrointestinal disorders) | 0 | 4
Dysphagia (Gastrointestinal disorders) | 0 | 4
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 | 5
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Lip pain (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 2 | 8
Nausea (Gastrointestinal disorders) | 29 | 23
Oral dysesthesia (Gastrointestinal disorders) | 1 | 1
Oral hemorrhage (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 3 | 2
Rectal hemorrhage (Gastrointestinal disorders) | 2 | 0
Rectal pain (Gastrointestinal disorders) | 3 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Stomach pain (Gastrointestinal disorders) | 2 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 7 | 3
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 5 | 0
Chills (General disorders and administration site conditions) | 3 | 1
Edema face (General disorders and administration site conditions) | 2 | 0
Edema limbs (General disorders and administration site conditions) | 18 | 18
Fatigue (General disorders and administration site conditions) | 49 | 50
Fever (General disorders and administration site conditions) | 1 | 3
Flu like symptoms (General disorders and administration site conditions) | 1 | 4
Infusion related reaction (General disorders and administration site conditions) | 25 | 1
Localized edema (General disorders and administration site conditions) | 4 | 3
Multi-organ failure (General disorders and administration site conditions) | 0 | 1
Non-cardiac chest pain (General disorders and administration site conditions) | 0 | 1
Pain (General disorders and administration site conditions) | 2 | 4
Gallbladder pain (Hepatobiliary disorders) | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 1
Immune system disorders - Other, specify (Immune system disorders) | 3 | 1
Eye infection (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 4 | 7
Meningitis (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 0 | 1
Papulopustular rash (Infections and infestations) | 1 | 0
Rhinitis infective (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 2 | 0
Skin infection (Infections and infestations) | 2 | 2
Tooth infection (Infections and infestations) | 1 | 0
Upper respiratory infection (Infections and infestations) | 5 | 8
Urinary tract infection (Infections and infestations) | 2 | 2
Infections and infestations - Other, specify (Infections and infestations) | 8 | 7
Bruising (Injury, poisoning and procedural complications) | 0 | 1
Burn (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 6 | 5
Fracture (Injury, poisoning and procedural complications) | 1 | 2
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 41 | 57
Alkaline phosphatase increased (Investigations) | 38 | 38
Aspartate aminotransferase increased (Investigations) | 34 | 49
Blood bilirubin increased (Investigations) | 1 | 0
Blood corticotrophin decreased (Investigations) | 0 | 1
Cholesterol high (Investigations) | 3 | 4
Creatinine increased (Investigations) | 37 | 25
Neutrophil count decreased (Investigations) | 34 | 26
Platelet count decreased (Investigations) | 46 | 44
Urine output decreased (Investigations) | 1 | 0
Weight gain (Investigations) | 1 | 1
Weight loss (Investigations) | 1 | 3
White blood cell decreased (Investigations) | 64 | 23
Investigations - Other, specify (Investigations) | 4 | 3
Anorexia (Metabolism and nutrition disorders) | 8 | 15
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 6 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 5 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 13 | 8
Hyponatremia (Metabolism and nutrition disorders) | 5 | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 2
Iron overload (Metabolism and nutrition disorders) | 2 | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 7
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 2 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6 | 3
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 3 | 3
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 9
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 7
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 2
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Cognitive disturbance (Nervous system disorders) | 1 | 0
Concentration impairment (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 5 | 4
Dysarthria (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 10 | 11
Extrapyramidal disorder (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 8 | 14
Intracranial hemorrhage (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 11 | 9
Tremor (Nervous system disorders) | 4 | 1
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 3 | 7
Confusion (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 4 | 4
Insomnia (Psychiatric disorders) | 8 | 6
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 | 3
Chronic kidney disease (Renal and urinary disorders) | 2 | 1
Urinary frequency (Renal and urinary disorders) | 2 | 3
Urinary incontinence (Renal and urinary disorders) | 2 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 1
Breast pain (Reproductive system and breast disorders) | 1 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 1 | 0
Scrotal pain (Reproductive system and breast disorders) | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0
Vaginal dryness (Reproductive system and breast disorders) | 3 | 1
Vaginal pain (Reproductive system and breast disorders) | 1 | 0
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 13
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 21 | 17
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 11 | 14
Erythroderma (Skin and subcutaneous tissue disorders) | 1 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 1
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 12
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 23 | 18
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 5 | 9
Hot flashes (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 21 | 18
Hypotension (Vascular disorders) | 1 | 2
Lymphedema (Vascular disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 1
Vascular disorders - Other, specify (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT02867384/Prot_SAP_000.pdf